CLINICAL TRIAL: NCT02910232
Title: In Vivo Clinical Trial of Porous Starch - Hydroxyapatite Composite Biomaterials for Bone Regeneration
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Sittiporn Punyanitya, Principal Investigator, Chiang Mai University
Other Study IDs: 0425/58
Record Dates: First submitted 2016-08-31; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Open Fracture of Foot
Keywords: Rice starch; Porous composite; Biomaterial; Bone regeneration; Clinical trial; Hydroxyapatite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: The groups were orthopedic patients and neurosurgical patients. The samples to fill the voiding space of bone and skull same as autografts.
  Interventions: Device: bone void filler

INTERVENTIONS:
Device: bone void filler — Bone void filler device prepared from porous starch-hydroxyapatite composites for bone regeneration

SUMMARY:
Biodegradable scaffold is an accepted and commercialized medical alternative choice for bone regeneration. In this project we will used our new invention, porous starch- hydroxyapatite composite, for in vivo clinical trial.

DETAILED DESCRIPTION:
The products were prepared from medical grade Thai rice starch mixed with high purity (>97%) hydroxyapatite powder from fresh cow bone, and already passed in vivo animal biocompatility test, then processed by freeze-drying. There were 44 volunteers from orthopedic and neurosurgical division, 4 and 40 patients, respectively.

ELIGIBILITY:
Inclusion Criteria:

* A patient who requires treatment by surgery and product implant in bone.
* Not indicate sex type
* 18-65 years
* Patients accepted participate in the study.
* Type of surgery will be treat for only bone.

Exclusion Criteria:

* Refused to join the study.
* Patients have an allergic history of carbohydrates and bovine bone.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There were 44 volunteers from orthopedic and neurosurgical division.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bone voids repairing | 6 months
  The primary outcome will be assessed from satisfactory grading by operative nurses and surgeons. Add a convenient storage, package removal, contamination risk, unused material disposal, size appropriateness, tolerability by hand, ease to cut, stability when wet, weight, and disturbance to operative field.

SECONDARY OUTCOMES:
Bone voids repairing | 6 months
  The short and long term safety and efficacy were assessed during real time operation, such as material dislodgement. Add a during follow up time for at least 1 months such as infection and allergic reaction by X-ray follow up assessment at 1, 3 and 6 months intervals, after operations.

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Materials and Ceramic Industrial Research Unit, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
yes, we plan

REFERENCES:
- [Result] Holzapfel BM, Reichert JC, Schantz JT, Gbureck U, Rackwitz L, Noth U, Jakob F, Rudert M, Groll J, Hutmacher DW. How smart do biomaterials need to be? A translational science and clinical point of view. Adv Drug Deliv Rev. 2013 Apr;65(4):581-603. doi: 10.1016/j.addr.2012.07.009. Epub 2012 Jul 20. PMID 22820527
- [Result] Dimitriou R, Jones E, McGonagle D, Giannoudis PV. Bone regeneration: current concepts and future directions. BMC Med. 2011 May 31;9:66. doi: 10.1186/1741-7015-9-66. PMID 21627784
- [Result] Mendes SC, Reis RL, Bovell YP, Cunha AM, van Blitterswijk CA, de Bruijn JD. Biocompatibility testing of novel starch-based materials with potential application in orthopaedic surgery: a preliminary study. Biomaterials. 2001 Jul;22(14):2057-64. doi: 10.1016/s0142-9612(00)00395-1. PMID 11426886
- See also: Accessed 29 June 2016 — http://www.marketsandmarkets.com/pdfdownload.asp?id=728